CLINICAL TRIAL: NCT02907450
Title: TolTwiCare : Qualitative Evaluation Routine Care From Primary Tolerance of a Prefabricated and Removable Orthosis
Acronym: TolTwiCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD/11/2-W; 2011-A01106-35 (Other: ANSM)
Record Dates: First submitted 2016-09-09; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Dentofacial Functional Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clinical evaluation of the tolerance of the orthosis (Experimental)
  Interventions: Device: TwiCare®.

INTERVENTIONS:
Device: TwiCare®.

SUMMARY:
The TwiCare® device is a removable brace that can be used in orthopedic referred to stimulate mandibular growth or in interception / contention.

The proposed research project will focus initially on assessing the comfort and safety of TwiCare® device. The orthopedic efficiency therefore not part of this study.

The comfort and safety of the brace will be evaluated firstly by the practitioner during the visit control around 2 ½ months (or 11 weeks) after the start of the port of the device, and with the help of a questionnaire completed by the patient at home 3 weeks and 6 weeks after the start of the port of the device, and during the control visit at 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients, where the laying of a brace phase of interception or contention after dental-facial orthodontic treatment is indicated (an intended age range of 8-18 years, not exhaustive or limiting) , recipient of a social security scheme, for which a management of the orthosis is acquired.
* incisor width compatible with the sizes of TwiCare® orthotics available, according to manufacturer's recommendations
* patient in good general health
* parent or guardian able to receive clear information, and express their opposition not to the patient's participation in this research
* for patients with malocclusions, the incisors (maxillary and mandibular) should be aligned.

Exclusion Criteria:

* General chronic health problem, unbalanced
* obvious oral ventilation
* history of temporomandibular dysfunction
* nocturnal episodes of severe bruxism
* unbalanced periodontal disease
* allergies or intolerances known to one of the constituents of the orthosis
* opposition of representatives of the parental authority (parent or guardian) or the patient himself at the patient's participation in this research
* patient unable to respond to the questionnaire
* monitoring difficulties (going on holiday, imminent change, remoteness, lack of motivation)
* simultaneous participation in intervention research
* pregnant Patient on examination of the latter, according to his age
* Incisive (maxilla and / or mandible) unaligned

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
No appearance of more than one injury that can not be attributed to causes other than the orthosis | 11 weeks

SECONDARY OUTCOMES:
The clinical evaluation of the compliance of the orthosis (occurrence of tooth movement, state of the brace, usual patient interview) | 11 weeks
The subjective assessment of the compliance of wearing the brace by patient by self questionnaire | 11 weeks
The subjective assessment of patient acceptability questionnaires self treatment | 11 weeks
The support type envisaged endline by the doctor | 11 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes -Service d'Odontologie Restauratrice et Chirurgicale, Nantes, France

IPD SHARING:
Plan to Share IPD: No